CLINICAL TRIAL: NCT05682261
Title: The Effect of Multiple Micronutrient Supplements in Reducing Anemia Among Women of Reproductive Age Compared to Iron-folic Acid at Kebribeyah District in Somali Regional State, Ethiopia- A Community-based Individual Randomized Control Trial
Brief Title: The Effect of Multiple Micronutrient Supplements in Reducing Anemia in Women of Reproductive Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethiopian Public Health Institute (Other Government)
Collaborators: Oklahoma State University (Other); Addis Ababa University (Other)
Responsible Party: Principal Investigator, Desalegn Kuche, Researcher for nutrition, Ethiopian Public Health Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EPHI_IRB_410_2021_2
Record Dates: First submitted 2022-12-04; First posted 2023-01-12 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2023-09

CONDITIONS: Anemia
Keywords: Multiple Micronutrient Supplements; Iron-folic acid; Anemia; Hemoglobin; Women of reproductive age
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Intervention Model Description: The three arms included in this trial are the multiple micronutrient supplement arm, iron-folic acid arm, and the placebo arm. This trial is a parallel-group community-based individual randomized control trial. The participants will be allocated randomly to the three arms and receive only the intervention assigned to them.
Who Masked: Participant, Outcomes Assessor
Masking Description: In the current trial, the outcome assessors and study subjects will both be blinded. The supplements being administered to participants, as well as who is in the intervention group and who is in the control group, will be masked from the assessors. The trial participants will be blinded to the kind of supplements being administered to them and the group to which they were assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Multiple micronutrient supplement arm (Experimental): The participants in this arm will receive United Nations International Multiple Micronutrient-Multiple Micronutrient Supplements. The recommended doses of UNIMMAP-MMS are vitamin A as retinol acetate (800 µg RAE), vitamin D as cholecalciferol (5 µg), vitamin E as alpha-tocopherol succinate (10 mg), vitamin C as ascorbic acid (70 mg), vitamin B1 as thiamin mononitrate (1.4 mg), vitamin B2 as riboflavin (1.4 mg), vitamin B3 as nicotinamide (18 mg), vitamin B6 as pyridoxine hydrochloride (1.9 mg), vitamin B12 as cyanocobalamin (2.6 µg), folic acid (680 µg), iron as ferrous fumarate (30 mg), zinc as zinc oxide (15 mg), copper as copper oxide (2 mg), selenium as sodium selenite (65 µg), iodine as potassium iodide (150 µg). The UNIMMAP-MMS in the tablet form will be used. We will give the supplementation twice a week and follow the study participants for 17 weeks.
  Interventions: Dietary Supplement: UNIMMAP-MMS
- Iron-folic acid supplement arm (Experimental): The participants in this arm will receive Iron-Folic Acid (IFA) supplements. The recommended doses of iron-folic acid are 30-60 mg of elemental iron and 400 µg of folic acid combined. In this trial, we will use ferrous sulfate with 30 mg of iron and 400 µg of folic acid in the form of capsule. The supplementation will be given to the study subjects twice a week for 17 weeks.
  Interventions: Dietary Supplement: IFA
- Control arm (Placebo Comparator): The participants in this arm will receive placebos made of sugar (lactose anhydrous). There is no active ingredient in the placebos. The placebos are lactose powder filled in the capsule. We will give placebos twice a week and will follow the study subjects for 17 weeks. The study subjects in this arm will be compensated with UNIMMAP-MMS at the end of the intervention.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: UNIMMAP-MMS — The study participants in this arm will receive the United Nations International Multiple Micronutrient Antenatal Preparation-Multiple Micronutrient Supplements (UNIMMAP-MMS) containing 15 micronutrients including 30 mg of iron and 400 µg of folic acid.
  Arms: Multiple micronutrient supplement arm
Dietary Supplement: IFA — The study participants in this arm will receive iron-folic acid supplements with 30 mg of iron and 400 µg of folic acid.
  Arms: Iron-folic acid supplement arm
Other: Placebo — The study participants in this arm will receive placebo made of sugar (lactose anhydrous).
  Arms: Control arm

SUMMARY:
The goal of this clinical trial is to test the effect of multiple micronutrient supplements in reducing anemia in women of reproductive age in comparison with iron-folic acid.

The main questions it aims to answer are:

* What is the effect of multiple micronutrient supplements in reducing anemia among women of reproductive age in comparison with iron-folic acid?
* What is the effect of multiple micronutrient supplements in reducing iron deficiency among women of reproductive age in comparison with iron-folic acid?

Participants will

* be given multiple micronutrient supplements, iron folic acid, or placebo twice weekly for 17 weeks
* be asked to respond to the interview
* provide blood, urine, and stool samples

Researchers will compare the control group with the intervention groups to see the effect of multiple micronutrient supplements on iron deficiency and anemia reduction.

DETAILED DESCRIPTION:
Women in developing countries are often at risk of micronutrient deficiencies due to inadequate micronutrient intake. Since various micronutrient deficiencies co-exist, multiple micronutrient supplements are recommended to combat their deficiencies. The purpose of this study is to assess the effects of multiple micronutrient supplements among women of reproductive age in reducing anemia compared with iron-folic acid as currently practiced in Ethiopia. The current study is a community-based individual randomized placebo-controlled trial. The trial is double blinded with three parallel groups. This trial will be conducted in three randomly selected kebeles (villages) in the Kebribeyah district in the Somali regional state. The sample size determined for this study is 305. There will be two intervention arms and one control arm in this trial. A third of participants will be in each arms. The intervention arms will will be supplemented with United Nations International Multiple Micronutrient Antenatal Preparation-Multiple Micronutrient Supplements (UNIMMAP-MMS) or iron-folic acid (IFA) and the control arm with placebos twice a week. The investigators will follow the study participants for 17 weeks. The primary outcome is a change in mean hemoglobin concentrations and reduction in anemia prevalence. Stratified randomization will be used to assign the participants randomly to the study arms. In the current trial, the outcome assessors and study subjects will both be blinded. The supplements being administered to participants, as well as who is in the intervention group and who is in the control group, will be masked from the assessors. The trial participants will be blinded to the kind of supplements being administered to them or the group to which they were assigned. The allocation sequence of participants will be concealed from the researcher who will assign the participants to the study arms. When the eligible woman meets the screening criteria and gives informed consent, she will be assigned an envelope that contains an allocation sequence. As outcome measures, the investigators will assess the reduction in overall anemia and iron deficiency anemia attributable to the supplementation. In addition, a complete blood count (CBC) will be tested for all study participants.

ELIGIBILITY:
Inclusion Criteria:

* Age range of 18-49 years.
* Mildly anemic (Hb=11.0-11.9 g/dl) or moderately anemic (Hb=8.0-10.9 g/dl) woman
* Permanent residents (lived for at least six months in the enumeration area)

Exclusion Criteria:

* A woman whose age is below or above the age range 18-49 year
* A pregnant woman
* Severely ill and incapacitated woman
* Non-permanent resident in the enumeration area
* Severely anemic (Hb <8.0 g/dl) woman
* A woman with Hb ≥12 g/dl

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The participants are expected to have the same gender identity as their biological sex.
Enrollment: 265 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2023-10-17 (Actual)

PRIMARY OUTCOMES:
Change in mean hemoglobin concentrations among women of reproductive age | Blood sample will be collected once at baseline and once at end-line in four months
  Hemoglobin concentration is measured in gram/deciliter from whole blood samples collected at baseline and end-line.
Change in overall anemia among women of reproductive age | Blood sample will be collected once at baseline and once at end-line in four months
  Anemia diagnosed when hemoglobin concentration test result is less than 12 g/dl

SECONDARY OUTCOMES:
Change in mean ferritin concentration among women of reproductive age | The serum samples will be collected once at the baseline and once at the end-line in four months
  Ferritin concentration is measured from serum ferritin in µg/L.
Change in iron deficiency anemia among women of reproductive age | Blood sample will be collected once at baseline and once at end-line in four months
  Iron deficiency anemia is diagnosed when hemoglobin concentration test result is less than 12 g/dl and the ferritin concentration test result is less than 15 µg/L

CONTACTS AND LOCATIONS:
Overall Officials: Masresha Tessema, PhD, Study Director — Ethiopian Public Health Institute (EPHI)
Locations (1):
- Ethiopian Public Health Institute, Addis Ababa, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: No
We do not currently have any plans to provide access to individual participant data. We may share the data once the key findings have been published. In addition, we need to obtain approval from the officials of the Ethiopian Public Health Institute.

REFERENCES:
- [Background] Chaparro CM, Suchdev PS. Anemia epidemiology, pathophysiology, and etiology in low- and middle-income countries. Ann N Y Acad Sci. 2019 Aug;1450(1):15-31. doi: 10.1111/nyas.14092. Epub 2019 Apr 22. PMID 31008520
- [Background] Ahmed F, Khan MR, Akhtaruzzaman M, Karim R, Marks GC, Banu CP, Nahar B, Williams G. Efficacy of twice-weekly multiple micronutrient supplementation for improving the hemoglobin and micronutrient status of anemic adolescent schoolgirls in Bangladesh. Am J Clin Nutr. 2005 Oct;82(4):829-35. doi: 10.1093/ajcn/82.4.829. PMID 16210713
- [Background] Gebreegziabher T, Stoecker BJ. Iron deficiency was not the major cause of anemia in rural women of reproductive age in Sidama zone, southern Ethiopia: A cross-sectional study. PLoS One. 2017 Sep 12;12(9):e0184742. doi: 10.1371/journal.pone.0184742. eCollection 2017. PMID 28898272
- [Background] Kassebaum NJ; GBD 2013 Anemia Collaborators. The Global Burden of Anemia. Hematol Oncol Clin North Am. 2016 Apr;30(2):247-308. doi: 10.1016/j.hoc.2015.11.002. PMID 27040955
- [Background] Multiple Micronutrient Supplement Technical Advisory Group (MMS-TAG); Micronutrient Forum (MNF). Expert consensus on an open-access United Nations International Multiple Micronutrient Antenatal Preparation-multiple micronutrient supplement product specification. Ann N Y Acad Sci. 2020 Jun;1470(1):3-13. doi: 10.1111/nyas.14322. Epub 2020 Mar 9. PMID 32153024
- [Background] Petry N, Olofin I, Hurrell RF, Boy E, Wirth JP, Moursi M, Donahue Angel M, Rohner F. The Proportion of Anemia Associated with Iron Deficiency in Low, Medium, and High Human Development Index Countries: A Systematic Analysis of National Surveys. Nutrients. 2016 Nov 2;8(11):693. doi: 10.3390/nu8110693. PMID 27827838
- [Background] Gomes F, Agustina R, Black RE, Christian P, Dewey KG, Kraemer K, Shankar AH, Smith ER, Thorne-Lyman A, Tumilowicz A, Bourassa MW. Multiple micronutrient supplements versus iron-folic acid supplements and maternal anemia outcomes: an iron dose analysis. Ann N Y Acad Sci. 2022 Jun;1512(1):114-125. doi: 10.1111/nyas.14756. Epub 2022 Feb 25. PMID 35218047
- [Derived] Kuche D, Abebe Z, Tessema M, Girma M, Hussen A, Baye K, Stoecker BJ. The effect of UNIMMAP multiple micronutrient supplements versus iron-folic acid and placebo in anemia reduction among women of reproductive age in Kebribeyah Woreda, Somali Regional State, Ethiopia: a study protocol for a community-based individual RCT. Trials. 2024 Mar 6;25(1):170. doi: 10.1186/s13063-024-08024-w. PMID 38448918